CLINICAL TRIAL: NCT04310774
Title: Concurrent Chemoradiotherapy Followed by Tegafur, Gimeracil and Oteracil Potassium Consolidation Chemotherapy in Patients With Locally Advanced Cervical Cancer: a Single Institute, Prospective, Single-arm Trial
Brief Title: CCRT Followed by Tegafur, Gimeracil and Oteracil Potassium in Cervical Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-S1
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Cervical Cancer; Chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Tegafur; gimeracil; potassium oxonate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consolidation therapy (Experimental): CCRT followed by Tegafur, Gimeracil and Oteracil Potassium Capsules consolidation chemotherapy
  Interventions: Drug: Tegafur, Gimeracil and Oteracil Potassium Capsules (one drug)

INTERVENTIONS:
Drug: Tegafur, Gimeracil and Oteracil Potassium Capsules (one drug) — CCRT followed by Tegafur, Gimeracil and Oteracil Potassium Capsules consolidation chemotherapy
  Other Names: CCRT followed by consolidation therapy

SUMMARY:
This is a single institute, single-arm, interventional trial to evaluate the efficacy and toxicity of concurrent chemoradiotherapy (CCRT) followed by Tegafur, Gimeracil and Oteracil Potassium Capsules consolidation chemotherapy in patients with locally advanced cervical cancer.

DETAILED DESCRIPTION:
This is a single institute, single-arm, interventional trial to evaluate the efficacy and toxicity of concurrent chemoradiotherapy (CCRT) followed by Tegafur, Gimeracil and Oteracil Potassium Capsules consolidation chemotherapy in patients with locally advanced cervical cancer. The main inclusive criteria are as follows: histology confirmed cervical cancer; 18-70 years old; 2018 International Federation of Gynecology and Obstetrics (FIGO) stage IIB-IIIC2; ECOG score <=1 point. The estimated enrollment is 200 patients. After enrollment, patients will receive CCRT, including external beam radiotherapy, intracavitary brachytherapy and concurrent chemotherapy. One month after the completion of CCRT, patients will receive 6 cycles of Tegafur, Gimeracil and Oteracil Potassium Capsules consolidation chemotherapy. The primary endpoint is progression free survival. And the secondary endpoints include overall survival, distant metastasis-free survival, local regional recurrence-free survival, acute toxicities, late toxicities, and treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

Histology confirmed cervical cancer; 18-70 years old; 2018 International Federation of Gynecology and Obstetrics (FIGO) stage IIB-IIIC2; Eastern Cooperative Oncology Group (ECOG) score <=1 point.; Adequate marrow: neutrophile granulocyte count ≥1.5*10^9/L, hemoglobin ≥ 80 g/L, platelet count ≥100*10^9/L; Normal liver and kidney function: Creatinine (Cr) < 1.5 mg/dl, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 2*upper limit of normal (ULN).

Exclusion Criteria:

Prior surgery (including pelvic or para-aortic lymph nodes resection, except for tumor biopsy), radiotherapy or chemotherapy to primary tumor or nodes; Prior malignancy;History of previous radiotherapy to the abdomen or pelvis; Pregnancy or lactation; Active infection with fever; Ssevere disease which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control, and emotional disturbance.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3-year/5-year
  The time from enrollment to disease progression or death from any cause, whichever is first

SECONDARY OUTCOMES:
Distant metastasis-free survival | 3-year/5-year
  The time from enrollment to distant metastasis or death from any cause, whichever is first.
Local regional recurrence-free survival | 3-year/5-year
  The time from enrollment to local regional recurrence or death from any cause, whichever is first.
Acute toxicities | From the start of treatment to 3 months
  Evaluated with CTCAE 5.0
Late toxicities | 3-year/5-year
  Evaluated with Radiation Therapy Oncology Group (RTOG)/EORTC late radiation morbidity scoring scheme

CONTACTS AND LOCATIONS:
Overall Officials: Ke Hu, MD, Study Chair — Radiotherapy department, Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No